CLINICAL TRIAL: NCT01612403
Title: Study the Effect of Oral Zinc Supplementation on High Molecular Weight Zinc Binding Protein in Semen
Acronym: supplement
Status: Completed | Type: Observational
Sponsor: mahmoud hussein hadwan (Other)
Responsible Party: Sponsor-Investigator, mahmoud hussein hadwan, Researcher, Babylon University
Organization: Babylon University (Other)
Other Study IDs: babil-1
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Asthenozoospermia
Keywords: zinc binding protein
MeSH Terms: conditions — Asthenozoospermia | interventions — Zinc Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single group: Single group: all participants receive same intervention throughout study (Non-randomised)
  Interventions: Dietary Supplement: zinc sulfate

INTERVENTIONS:
Dietary Supplement: zinc sulfate — every participant took two capsules of zinc sulfate per day for three months (each one 220mg)
  Other Names: infertility

SUMMARY:
There are several causes leading to male infertility, like oxidative stress, and nutritional deficiency of trace elements like zinc. Zinc in human seminal plasma was divided into three types of ligands which are high (HMW), intermediate (IMW), and low molecular weight ligands (LMW). The present study was conducted to study the effect of Zn supplementation on the quantitative and qualitative characteristics of semen along with Zinc Binding Protein levels in semen of patients with asthenozoospmia.

DETAILED DESCRIPTION:
Elevation of ROS levels lead to an increase the oxidation of HMW-Zn binding proteins in seminal plasma of asthenozoospermic subjects. Zinc supplementation restores HMW-Zn% in seminal plasma of asthenozoospermic subjects to normal value. LMW-Zn% is elevated in seminal plasma of asthenozoospermic patients. It may be because increment the levels of semenogelin in seminal plasma of asthenozoospermic subjects. Zinc supplementation elevates LMW-Zn% in seminal plasma of asthenozoospermic subjects to more than normal value, this may be because of its enhancement of the synthesis of metallothioneins (Low molecular weight zinc binding protein).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were the presence of asthenozoospermia in the semen sample.

Exclusion Criteria:

* the absence of endocrinopathy,
* varicocele, and
* female factor infertility. Smokers and alcoholic men were excluded from the study because of their recognized high seminal ROS levels and decreased antioxidant levels.

Ages: 27 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes 37 subfertile male partners from couples who had consulted the infertility clinic of the Babil hospital of maternity (Hilla city/ IRAQ).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
high molecular weight zinc binding protein | at the end of three months
  elevated levels of high molecular weight zinc binding protein to normal value

SECONDARY OUTCOMES:
qualitative semen parameters | at the end of three months
  Volume of semen, progressive sperm motility percentage and total normal sperm count increased after zinc sulfate supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud H. hadwan, Dr., Principal Investigator — babylon university / Iraq
Locations (2):
- Iraq (2):
  - Babylon university/ college of science, Hillah, Hilla
  - Babylon University, Hillah, Hilla

REFERENCES:
- [Derived] Hadwan MH, Almashhedy LA, Alsalman AR. Oral zinc supplementation restores high molecular weight seminal zinc binding protein to normal value in Iraqi infertile men. BMC Urol. 2012 Nov 13;12:32. doi: 10.1186/1471-2490-12-32. PMID 23145537